CLINICAL TRIAL: NCT01505634
Title: A Phase II, Randomized, Active Comparator-Controlled Clinical Trial to Study the Safety, Tolerability, and Efficacy of MK-7655 + Imipenem/Cilastatin Versus Imipenem/Cilastatin Alone in Patients With Complicated Urinary Tract Infection (cUTI)
Brief Title: Safety, Tolerability, and Efficacy of MK-7655 (Relebactam) + Imipenem/Cilastatin Versus Imipenem/Cilastatin Alone for Treating Complicated Urinary Tract Infection (cUTI) (MK-7655-003)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7655-003; 2011-005707-32 (EudraCT Number); MK-7655-003 (Other: Merck Protocol Number)
Record Dates: First submitted 2012-01-04; First posted 2012-01-06 (Estimated); Results first posted 2019-05-24 (Actual); Last update posted 2019-05-24 (Actual); Status verified 2019-04

CONDITIONS: Urinary Tract Infections; Pyelonephritis
Keywords: Relebactam; MK-7655; Imipenem; Urinary Tract Infections; Pyelonephritis; Urologic Diseases; beta-Lactamase Inhibitors; Anti-Bacterial and Anti-Infective Agent
MeSH Terms: conditions — Urinary Tract Infections; Pyelonephritis; Urologic Diseases | interventions — relebactam; Imipenem; Cilastatin; Cilastatin, Imipenem Drug Combination; Ciprofloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Relebactam 250 mg with imipenem/cilastatin (Experimental): Relebactam 250 mg IV co-administered with 500 mg of imipenem/cilastatin once every 6 hours for a minimum of 96 hours. After 96 hours of IV treatment, participants may be switched to 500 mg ciprofloxacin (as optional oral therapy following minimum duration of IV study drug), administered orally, twice daily for the remainder of the study. Antibiotic therapy (IV and oral combined) should not exceed 14 days.
  Interventions: Drug: Relebactam 250 mg; Drug: imipenem/cilastatin 500 mg; Drug: Ciprofloxacin
- Relebactam 125 mg with imipenem/cilastatin (Experimental): Relebactam 125 mg IV co-administered with 500 mg of imipenem/cilastatin once every 6 hours for a minimum of 96 hours. After 96 hours of IV treatment, participants may be switched to 500 mg ciprofloxacin (as optional oral therapy following minimum duration of IV study drug), administered orally, twice daily for the remainder of the study. Antibiotic therapy (IV and oral combined) should not exceed 14 days.
  Interventions: Drug: Relebactam 125 mg; Drug: imipenem/cilastatin 500 mg; Drug: Ciprofloxacin
- Relebactam placebo with imipenem/cilastatin (Placebo Comparator): Matching placebo for relebactam (0.9% normal saline) IV co-administered with 500 mg dose of imipenem/cilastatin once every 6 hours for a minimum of 96 hours. After 96 hours of IV treatment, participants may be switched to 500 mg ciprofloxacin (as optional oral therapy following minimum duration of IV study drug), administered orally, twice daily for the remainder of the study. Antibiotic therapy (IV and oral combined) should not exceed 14 days.
  Interventions: Drug: imipenem/cilastatin 500 mg; Drug: Placebo to relebactam; Drug: Ciprofloxacin

INTERVENTIONS:
Drug: Relebactam 250 mg — Participants randomized to receive relebactam 250 mg will be administered a 250 mg dose of relebactam IV in a blinded fashion once every 6 hours with each dose infused over a 30-minute interval.
  Other Names: MK-7655
  Arms: Relebactam 250 mg with imipenem/cilastatin
Drug: Relebactam 125 mg — Participants randomized to receive relebactam 125 mg will be administered a 125 mg dose of relebactam IV in a blinded-treatment fashion once every 6 hours with each dose infused over a 30-minute interval.
  Other Names: MK-7655
  Arms: Relebactam 125 mg with imipenem/cilastatin
Drug: imipenem/cilastatin 500 mg — A 500 mg dose of imipenem/cilastatin will be administered IV in an open-label fashion once every 6 hours with each dose infused over a 30-minute interval.
  Other Names: PRIMAXIN®, TIENAM®
Drug: Placebo to relebactam — Participants randomized to receive imipenem/cilastatin alone will receive a placebo-matching infusion of IV normal saline (0.9%) once every 6 hours.
  Arms: Relebactam placebo with imipenem/cilastatin
Drug: Ciprofloxacin — After at least 96 hours of IV treatment, participants may be switched, at the discretion of the investigator, to 500 mg ciprofloxacin, administered orally, twice daily

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and tolerability of adding 125 mg or 250 mg doses of MK-7655 (relebactam) to imipenem/cilastatin in adults 18 years or older with complicated urinary tract infection (cUTI). The primary hypothesis is that the relebactam + imipenem/cilastatin treatment regimen is non-inferior to imipenem/cilastatin with respect to the proportion of participants with a favorable microbiological response at completion of intravenous (IV) study therapy.

ELIGIBILITY:
Inclusion Criteria:

- Clinically suspected and/or bacteriologically documented cUTI or acute

pyelonephritis judged by the investigator to be serious (requiring hospitalization and treatment with IV antibiotic therapy)

- Pyuria, determined by a midstream clean-catch (MSCC) or catheterized

(indwelling or straight catheter) urine specimen with greater than or equal to 10 white blood cells (WBCs) per high-power field (hpf) on standard examination of urine sediment or greater than or equal to 10 WBCs/mm3 in unspun urine

- One positive urine culture within 48 hours of enrollment

Exclusion Criteria:

- Complete obstruction of any portion of the urinary tract (requiring a

permanent indwelling urinary catheter or instrumentation), a known ileal loop, or intractable vesico-ureteral reflux

* A temporary indwelling urinary catheter is in place and cannot be removed at study entry.
* Perinephric or intrarenal abscess or known or suspected prostatitis
* Uncomplicated UTI
* Any history of recent accidental trauma to the pelvis or urinary tract
* Any amount of effective antibiotic therapy after obtaining the urine culture for admission to this study and prior to the administration of the first dose of IV study therapy
* An infection which has been treated with greater than 24 hours of systemic antibiotic therapy known to be effective against the presumed or documented etiologic pathogen(s) within the 72-hour period immediately prior to consideration for entry into the study
* History of serious allergy, hypersensitivity (e.g., anaphylaxis), or any

serious reaction to carbapenem antibiotics, any cephalosporins, penicillins, or other beta (β)-lactam agents

* History of serious allergy, hypersensitivity (e.g., anaphylaxis), or any serious reaction to other beta-lactam inhibitors (e.g., tazobactam, sulbactam, clavulanic acid)
* History of a seizure disorder
* Currently being treated with valproic acid or has received treatment with

valproic acid in the 2 weeks prior to screening.

* Rapidly progressive or terminal illness unlikely to survive the approximately 6 to 8 week study period
* Pregnant or expecting to conceive, breast feeding, or plans to breast feed

during the study

- A response to all study therapy (IV study therapy or subsequent oral

ciprofloxacin) within the timeframe of treatment specified in this protocol is

considered unlikely.

- Concurrent infection that would interfere with evaluation of response to

the study antibiotics

- Need for concomitant systemic antimicrobial agents in addition to those

designated in the various study treatment groups (use of vancomycin, daptomycin, or linezolid is allowed for certain infections)

* cUTI due to a confirmed fungal pathogen
* Currently receiving immunosuppressive therapy, including use of high-dose

corticosteroids

* Prior recipient of a renal transplantation
* Laboratory abnormalities as specified in protocol
* History of any other illness that, in the opinion of the investigator, might

confound the results of the study or pose additional risk in administering the study drug

- Currently participating in, or has participated in, any other clinical study

involving the administration of investigational or experimental medication (not

licensed by regulatory agencies) at the time of presentation or during the previous 30 days prior to screening or is anticipated to participate in such a clinical study during the course of this trial

- Estimated or actual creatinine clearance of <5 mL/minute, or is currently undergoing hemodialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2012-05-16 (Actual); Primary Completion 2015-07-28 (Actual); Study Completion 2015-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Sims M, Mariyanovski V, McLeroth P, Akers W, Lee YC, Brown ML, Du J, Pedley A, Kartsonis NA, Paschke A. Prospective, randomized, double-blind, Phase 2 dose-ranging study comparing efficacy and safety of imipenem/cilastatin plus relebactam with imipenem/cilastatin alone in patients with complicated urinary tract infections. J Antimicrob Chemother. 2017 Sep 1;72(9):2616-2626. doi: 10.1093/jac/dkx139. PMID 28575389

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled with complicated urinary tract infection (cUTI) or acute pyelonephritis judged by the investigator to be serious (requiring hospitalization and intravenous (IV) antibiotic therapy); pyuria; and 1 positive urine culture within 48 hours of enrollment.
Period: Overall Study
Arm/Group | Relebactam 250 mg With Imipenem/Cilastatin | Relebactam 125 mg With Imipenem/Cilastatin | Relebactam Placebo With Imipenem/Cilastatin
Started | 101 | 101 | 100
Treated | 99 | 99 | 100
Completed | 92 | 91 | 94
Not Completed | 9 | 10 | 6
Not completed — Withdrawal by Subject | 2 | 5 | 1
Not completed — Physician Decision | 1 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Insufficient supply of drug at site | 1 | 0 | 0
Not completed — Protocol Violation | 2 | 0 | 0
Not completed — Lost to Follow-up | 1 | 4 | 4
Not completed — Death | 1 | 0 | 0
Not completed — In a conflict zone | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Relebactam 250 mg With Imipenem/Cilastatin | Relebactam 125 mg With Imipenem/Cilastatin | Relebactam Placebo With Imipenem/Cilastatin | Total
Number analyzed (Participants) | 101 | 101 | 100 | 302
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.9 (17.3) | 55.9 (17.5) | 55.7 (19.2) | 56.5 (18.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 60 | 42 | 153
  Male | 50 | 41 | 58 | 149

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Favorable Microbiological Response at Completion of IV Study Therapy
Description: Microbiological response (MR) was assessed based on results of bacterial cultures obtained at completion of IV study medication relative to cultures obtained at baseline. A favorable microbiological response was defined as eradication of all pathogens identified at baseline. Microbiological response was assessed separately for each participant and pathogen identified in the Microbiologically Evaluable (ME) population that included participants with a urine culture confirmed to be positive for at least 1 gram-negative and/or anaerobic pathogen(s) commonly isolated in UTI. The overall microbiological response was determined as "favorable" if all pathogens isolated from a participant at baseline demonstrated a "favorable" response (eradication) at the time point evaluated.
Time Frame: At time of last IV dose of study drug (up to post-randomization day 14)
Population: All participants in the ME population with non-missing/non-indeterminate response.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Relebactam 250 mg With Imipenem/Cilastatin | Relebactam 125 mg With Imipenem/Cilastatin | Relebactam Placebo With Imipenem/Cilastatin
Number analyzed (Participants) | 67 | 71 | 75
Percentage of Participants | 95.5 [87.5 to 99.1] | 98.6 [92.4 to 100.0] | 98.7 [92.8 to 100.0]
Statistical Analysis 1: Comparison: Relebactam 250 mg With Imipenem/Cilastatin vs Relebactam Placebo With Imipenem/Cilastatin; Percent Difference (Diff) in Favorable MR; Test type: Non-Inferiority — Non-inferiority for the relebactam 250 mg + imipenem/cilastatin group versus the Placebo for relebactam + imipenem/cilastatin group was demonstrated if the lower bound of the 95% CI was not lower than the pre-specified non-inferiority margin of -15%; p = 0.005, Miettinen and Nurminen; Percent Difference = -3.1, 95% CI 2-sided [-11.2 to 3.2] — Relebactam minus Placebo
Statistical Analysis 2: Comparison: Relebactam 125 mg With Imipenem/Cilastatin vs Relebactam Placebo With Imipenem/Cilastatin; Percent Diff in Favorable MR; Test type: Non-Inferiority — Non-inferiority for the relebactam 125 mg + imipenem/cilastatin group versus the Placebo for relebactam + imipenem/cilastatin group was demonstrated if the lower bound of the 95% CI was not lower than the pre-specified non-inferiority margin of -15%; p < 0.001, Miettinen and Nurminen; Percent Difference = -0.1, 95% CI 2-sided [-6.4 to 5.9] — Relebactam minus Placebo

2. Primary Outcome: Percentage of Participants With an Elevated Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT) Laboratory Value That Was Greater Than or Equal to 5 Times the Upper Limit of Normal (ULN)
Description: All randomized participants who received ≥1 dose of study treatment had AST and ALT levels measured up to 14 days following completion of all study medication. Participants who had 2 confirmed elevations of either AST or ALT that were 5 times ULN or greater were recorded.
Time Frame: Up to 14 days following completion of all study therapy (up to 28 days)
Population: All randomized participants who received ≥ 1 dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Relebactam 250 mg With Imipenem/Cilastatin | Relebactam 125 mg With Imipenem/Cilastatin | Relebactam Placebo With Imipenem/Cilastatin
Number analyzed (Participants) | 99 | 99 | 100
Percentage of participants | 1.0 | 1.0 | 0
Statistical Analysis 1: Comparison: Relebactam 250 mg With Imipenem/Cilastatin vs Relebactam Placebo With Imipenem/Cilastatin; Percent Diff in Participants with Event of Clinical Interest (ECI) #1; Test type: Other — ECI #1 is a confirmed elevated AST or ALT ≥5X ULN. Inferential testing for statistical significance with p-values and 95% confidence intervals was performed to provide a comparison between the relebactam 250 mg + imipenem/cilastatin group versus the Placebo for relebactam + imipenem/cilastatin group; p = 0.315, Miettinen and Nurminen; Percent Difference = 1.0, 95% CI 2-sided [-2.7 to 5.5] — Relebactam minus Placebo
Statistical Analysis 2: Comparison: Relebactam 125 mg With Imipenem/Cilastatin vs Relebactam Placebo With Imipenem/Cilastatin; Percent Diff in Participants with ECI #1; Test type: Other — ECI #1 is a confirmed elevated AST or ALT ≥5X ULN. Inferential testing for statistical significance with p-values and 95% confidence intervals was performed to provide a comparison between the relebactam 125 mg + imipenem/cilastatin group versus the Placebo for relebactam + imipenem/cilastatin group; p = 0.315, Miettinen and Nurminen; Percent Difference = 1.0, 95% CI 2-sided [-2.7 to 5.5] — Relebactam minus Placebo

3. Primary Outcome: Percentage of Participants With Elevated AST or ALT Laboratory Values ≥ 3 Times the ULN, as Well as Elevated Total Bilirubin ≥ 2 Times the ULN, and Alkaline Phosphatase Values That Were < 2 Times the ULN
Description: All randomized participants who received ≥1 dose of study treatment had AST, ALT, total bilirubin, and Alkaline Phosphatase (ALP) levels measured up to 14 days following completion of all study medication. Participants who had elevations of AST or ALT that were ≥3 times ULN, total bilirubin measurements that were ≥2 times ULN and, at the same time, an ALP measurement of < 2X ULN were recorded.
Time Frame: Up to 14 days following completion of all study therapy (up to 28 days)
Population: All randomized participants who received ≥ 1 dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Relebactam 250 mg With Imipenem/Cilastatin | Relebactam 125 mg With Imipenem/Cilastatin | Relebactam Placebo With Imipenem/Cilastatin
Number analyzed (Participants) | 99 | 99 | 100
Percentage of participants | 0 | 0 | 0
Statistical Analysis 1: Comparison: Relebactam 250 mg With Imipenem/Cilastatin vs Relebactam Placebo With Imipenem/Cilastatin; Percent Diff Participants with ECI #2; Test type: Other — Event of Clinical Interest (ECI) #2 is elevated AST or ALT ≥3X ULN, elevated total bilirubin ≥2X ULN, and with an ALP <2X ULN. Inferential testing for statistical significance with p-values and 95% confidence intervals was performed to provide a comparison between the relebactam 250 mg + imipenem/cilastatin group versus the Placebo for relebactam + imipenem/cilastatin group; p > 0.999, Miettinen and Nurminen — No participants met the criteria for ECI #2; Percent Difference = 0.0, 95% CI 2-sided [-3.7 to 3.8] — Relebactam minus Placebo
Statistical Analysis 2: Comparison: Relebactam 125 mg With Imipenem/Cilastatin vs Relebactam Placebo With Imipenem/Cilastatin; Percent Diff in Participants with ECI #2; Test type: Other — Event of Clinical Interest (ECI) #2 is elevated AST or ALT ≥3X ULN, elevated total bilirubin ≥2X ULN, and with an ALP <2X ULN. Inferential testing for statistical significance with p-values and 95% confidence intervals was performed to provide a comparison between the relebactam 125 mg + imipenem/cilastatin group versus the Placebo for relebactam + imipenem/cilastatin group; p > 0.999, Miettinen and Nurminen — No participants met the criteria for ECI #2; Percent Difference = 0.0, 95% CI 2-sided [-3.7 to 3.8] — Relebactam minus Placebo

4. Primary Outcome: Percentage of Participants With at Least 1 Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product/protocol-specified procedure, whether or not considered related to the medicinal product/protocol-specified procedure. Any worsening of a preexisting condition temporally associated with the use of the product was also an AE.
Time Frame: Up to 14 days following completion of all study therapy (up to 28 days)
Population: All randomized participants who received ≥1 dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Relebactam 250 mg With Imipenem/Cilastatin | Relebactam 125 mg With Imipenem/Cilastatin | Relebactam Placebo With Imipenem/Cilastatin
Number analyzed (Participants) | 99 | 99 | 100
Percentage of participants | 28.3 | 29.3 | 30.0
Statistical Analysis 1: Comparison: Relebactam 250 mg With Imipenem/Cilastatin vs Relebactam Placebo With Imipenem/Cilastatin; Percent Diff in Participants with AEs; Test type: Other — Difference in percentage and 95% CI are based on unconditional and asymptotic Miettinen and Nurminen method; Percent Difference = -1.7, 95% CI [-14.3 to 10.9] — Relebactam minus Placebo
Statistical Analysis 2: Comparison: Relebactam 125 mg With Imipenem/Cilastatin vs Relebactam Placebo With Imipenem/Cilastatin; Percent Diff in Participants with AEs; Test type: Other — Difference in percentage and 95% CI are based on unconditional and asymptotic Miettinen and Nurminen method; Percent Difference = -0.7, 95% CI 2-sided [-13.4 to 12.0] — Relebactam minus Placebo

5. Primary Outcome: Percentage of Participants With Any Serious Adverse Event (SAE)
Description: A SAE was an AE that resulted in death, was life threatening, resulted in persistent or significant disability/incapacity, resulted in or prolonged an existing inpatient hospitalization, was a congenital anomaly/birth defect, was a cancer, was associated with an overdose, was another important medical event.
Time Frame: Up to 14 days following completion of all study therapy (up to 28 days)
Population: All randomized participants who received ≥1 dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Relebactam 250 mg With Imipenem/Cilastatin | Relebactam 125 mg With Imipenem/Cilastatin | Relebactam Placebo With Imipenem/Cilastatin
Number analyzed (Participants) | 99 | 99 | 100
Percentage of participants | 3.0 | 1.0 | 3.0
Statistical Analysis 1: Comparison: Relebactam 250 mg With Imipenem/Cilastatin vs Relebactam Placebo With Imipenem/Cilastatin; Percent Diff in Participants with SAEs; Test type: Other — Difference in percentage and 95% CI are based on unconditional and asymptotic Miettinen and Nurminen method; Percent Difference = 0.0, 95% CI 2-sided [-5.8 to 5.9] — Relebactam minus Placebo
Statistical Analysis 2: Comparison: Relebactam 125 mg With Imipenem/Cilastatin vs Relebactam Placebo With Imipenem/Cilastatin; Percent Diff in Participants with SAEs; Test type: Other — Difference in percentage and 95% CI are based on unconditional and asymptotic Miettinen and Nurminen method; Percent Difference = -2.0, 95% CI 2-sided [-7.6 to 2.8] — Relebactam minus Placebo

6. Primary Outcome: Percentage of Participants With Any Drug-related AE
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product/protocol-specified procedure, whether or not considered related to the medicinal product/protocol-specified procedure. Any worsening of a preexisting condition temporally associated with the use of the product was also an AE. A drug-related (DR) AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product that the investigator determined to be possibly, probably, or definitely related to the treatment.
Time Frame: Up to 14 days following completion of all study therapy (up to 28 days)
Population: All randomized participants who received ≥1 dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Relebactam 250 mg With Imipenem/Cilastatin | Relebactam 125 mg With Imipenem/Cilastatin | Relebactam Placebo With Imipenem/Cilastatin
Number analyzed (Participants) | 99 | 99 | 100
Percentage of participants | 10.1 | 9.1 | 9.0
Statistical Analysis 1: Comparison: Relebactam 250 mg With Imipenem/Cilastatin vs Relebactam Placebo With Imipenem/Cilastatin; Percent Diff in Participants with DR AEs; Test type: Other — Difference in percentage and 95% CI are based on unconditional and asymptotic Miettinen and Nurminen method; Percent Difference = 1.1, 95% CI 2-sided [-7.5 to 9.8] — Relebactam minus Placebo
Statistical Analysis 2: Comparison: Relebactam 125 mg With Imipenem/Cilastatin vs Relebactam Placebo With Imipenem/Cilastatin; Percent Diff in Participants with DR AEs; Test type: Other — Difference in percentage and 95% CI are based on unconditional and asymptotic Miettinen and Nurminen method; Percent Difference = 0.1, 95% CI 2-sided [-8.4 to 8.6] — Relebactam minus Placebo

7. Primary Outcome: Percentage of Participants With a Drug-related SAE
Description: A serious, drug-related (DR) AE was an AE that resulted in death, was life threatening, resulted in persistent or significant disability/incapacity, resulted in or prolonged an existing inpatient hospitalization, was a congenital anomaly/birth defect, was a cancer, was associated with an overdose, was another important medical event. The SAE was determined to be possibly, probably, or definitely related to the treatment by the investigator.
Time Frame: Up to 42 days following completion of all study therapy (up to 56 days)
Population: All randomized participants who received ≥1 dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Relebactam 250 mg With Imipenem/Cilastatin | Relebactam 125 mg With Imipenem/Cilastatin | Relebactam Placebo With Imipenem/Cilastatin
Number analyzed (Participants) | 99 | 99 | 100
Percentage of participants | 1.0 | 0 | 1.0
Statistical Analysis 1: Comparison: Relebactam 250 mg With Imipenem/Cilastatin vs Relebactam Placebo With Imipenem/Cilastatin; Percent Diff in Participants with DR SAEs; Test type: Other — Difference in percentage and 95% CI are based on unconditional and asymptotic Miettinen and Nurminen method; Percent Difference = 0.0, 95% CI 2-sided [-4.5 to 4.6] — Relebactam minus Placebo
Statistical Analysis 2: Comparison: Relebactam 125 mg With Imipenem/Cilastatin vs Relebactam Placebo With Imipenem/Cilastatin; Percent Diff in Participants with DR SAEs; Test type: Other — Difference in percentage and 95% CI are based on unconditional and asymptotic Miettinen and Nurminen method; Percent Difference = -1.0, 95% CI 2-sided [-5.5 to 2.8] — Relebactam minus Placebo

8. Primary Outcome: Percentage of Participants Who Discontinued IV Study Therapy Due to an AE
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product/protocol-specified procedure, whether or not considered related to the medicinal product/protocol-specified procedure. Any worsening of a pre-existing condition temporally associated with the use of the product was also an AE.
Time Frame: Up to 14 days
Population: All randomized participants who received ≥1 dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Relebactam 250 mg With Imipenem/Cilastatin | Relebactam 125 mg With Imipenem/Cilastatin | Relebactam Placebo With Imipenem/Cilastatin
Number analyzed (Participants) | 99 | 99 | 100
Percentage of participants | 3.0 | 1.0 | 2.0
Statistical Analysis 1: Comparison: Relebactam 250 mg With Imipenem/Cilastatin vs Relebactam Placebo With Imipenem/Cilastatin; Percent Diff in Participants with Discons Due to AEs; Test type: Other — Difference in percentage and 95% CI are based on unconditional and asymptotic Miettinen and Nurminen method; Percent Difference = 1.0, 95% CI 2-sided [-4.4 to 6.8] — Relebactam minus Placebo
Statistical Analysis 2: Comparison: Relebactam 125 mg With Imipenem/Cilastatin vs Relebactam Placebo With Imipenem/Cilastatin; Percent Diff in Participants with Discons Due to AEs; Test type: Other — Difference in percentage and 95% CI are based on unconditional and asymptotic Miettinen and Nurminen method; Percent Difference = -1.0, 95% CI 2-sided [-6.1 to 3.7] — Relebactam minus Placebo

9. Primary Outcome: Percentage of Participants Who Discontinued IV Study Therapy Due to a Drug-related AE
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product/protocol-specified procedure, whether or not considered related to the medicinal product/protocol-specified procedure. Any worsening of a preexisting condition temporally associated with the use of the product was also an AE. A drug-related AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product that the investigator determined to be possibly, probably, or definitely related to the treatment.
Time Frame: Up to 14 days
Population: All randomized participants who received ≥1 dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Relebactam 250 mg With Imipenem/Cilastatin | Relebactam 125 mg With Imipenem/Cilastatin | Relebactam Placebo With Imipenem/Cilastatin
Number analyzed (Participants) | 99 | 99 | 100
Percentage of participants | 2.0 | 1.0 | 1.0
Statistical Analysis 1: Comparison: Relebactam 250 mg With Imipenem/Cilastatin vs Relebactam Placebo With Imipenem/Cilastatin; Percent Diff in Participants with Discons Due to DR AEs; Test type: Other — Difference in percentage and 95% CI are based on unconditional and asymptotic Miettinen and Nurminen method; Percent Difference = 1.0, 95% CI 2-sided [-3.6 to 6.2] — Relebactam minus Placebo
Statistical Analysis 2: Comparison: Relebactam 125 mg With Imipenem/Cilastatin vs Relebactam Placebo With Imipenem/Cilastatin; Percent Diff in Participants with Discons Due to DR AEs; Test type: Other — Difference in percentage and 95% CI are based on unconditional and asymptotic Miettinen and Nurminen method; Percent Difference = 0.0, 95% CI 2-sided [-4.5 to 4.6] — Relebactam minus Placebo

10. Primary Outcome: Percentage of Participants With Specific AEs With Incidence of >= 4 Participants in One Treatment Group
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product/protocol-specified procedure, whether or not considered related to the medicinal product/protocol-specified procedure. Any worsening of a preexisting condition temporally associated with the use of the product was also an AE. Analysis includes specific adverse events with an incidence of ≥4 participants in one treatment group or system organ class.
Time Frame: Up to 14 days following completion of all study therapy (up to 28 days)
Population: All randomized participants who received ≥1 dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Relebactam 250 mg With Imipenem/Cilastatin | Relebactam 125 mg With Imipenem/Cilastatin | Relebactam Placebo With Imipenem/Cilastatin
Number analyzed (Participants) | 99 | 99 | 100
Percentage of participants
  Diarrhoea | 5.1 | 2.0 | 4.0
  Nausea | 4.0 | 6.1 | 4.0
  Bacteriuria | 1.0 | 2.0 | 4.0
  White blood cells urine positive | 1.0 | 1.0 | 4.0
  Headache | 7.1 | 3.0 | 4.0
Statistical Analysis 1: Comparison: Relebactam 250 mg With Imipenem/Cilastatin vs Relebactam Placebo With Imipenem/Cilastatin; Percent Diff in Participants with AEs with Rate ≥4: Diarrhoea; Test type: Other — Difference in percentage and 95% CI are based on unconditional and asymptotic Miettinen and Nurminen method; Percent Difference = 1.1, 95% CI 2-sided [-5.5 to 7.8] — Relebactam minus Placebo
Statistical Analysis 2: Comparison: Relebactam 125 mg With Imipenem/Cilastatin vs Relebactam Placebo With Imipenem/Cilastatin; Percent Diff in Participants with AEs with Rate ≥4: Diarrhoea; Test type: Other — Difference in percentage and 95% CI are based on unconditional and asymptotic Miettinen and Nurminen method; Percent Difference = -2.0, 95% CI 2-sided [-8.1 to 3.6] — Relebactam minus Placebo
Statistical Analysis 3: Comparison: Relebactam 250 mg With Imipenem/Cilastatin vs Relebactam Placebo With Imipenem/Cilastatin; Percent Diff in Participants with AEs with Rate ≥4: Nausea; Test type: Other — Difference in percentage and 95% CI are based on unconditional and asymptotic Miettinen and Nurminen method; Percent Difference = 0.0, 95% CI 2-sided [-6.4 to 6.5] — Relebactam minus Placebo
Statistical Analysis 4: Comparison: Relebactam 125 mg With Imipenem/Cilastatin vs Relebactam Placebo With Imipenem/Cilastatin; Percent Diff in Participants with AEs with Rate ≥4: Nausea; Test type: Other — Difference in percentage and 95% CI are based on unconditional and asymptotic Miettinen and Nurminen method; Percent Difference = 2.1, 95% CI 2-sided [-4.6 to 9.2] — Relebactam minus Placebo
Statistical Analysis 5: Comparison: Relebactam 250 mg With Imipenem/Cilastatin vs Relebactam Placebo With Imipenem/Cilastatin; Percent Diff in Participants with AEs with Rate ≥4: Bacteriuria; Test type: Other — Difference in percentage and 95% CI are based on unconditional and asymptotic Miettinen and Nurminen method; Percent Difference = -3.0, 95% CI 2-sided [-9.0 to 1.9] — Relebactam minus Placebo
Statistical Analysis 6: Comparison: Relebactam 125 mg With Imipenem/Cilastatin vs Relebactam Placebo With Imipenem/Cilastatin; Percent Diff in Participants with AEs with Rate ≥4: Bacteriuria; Test type: Other — Difference in percentage and 95% CI are based on unconditional and asymptotic Miettinen and Nurminen method; Percent Difference = -2.0, 95% CI 2-sided [-8.1 to 3.6] — Relebactam minus Placebo
Statistical Analysis 7: Comparison: Relebactam 250 mg With Imipenem/Cilastatin vs Relebactam Placebo With Imipenem/Cilastatin; Percent Diff in Participants with AEs with Rate ≥4: White blood cells urine positive; Test type: Other — Difference in percentage and 95% CI are based on unconditional and asymptotic Miettinen and Nurminen method; Percent Difference = -3.0, 95% CI 2-sided [-9.0 to 1.9] — Relebactam minus Placebo
Statistical Analysis 8: Comparison: Relebactam 125 mg With Imipenem/Cilastatin vs Relebactam Placebo With Imipenem/Cilastatin; Percent Diff in Participants with AEs with Rate ≥4: White blood cells urine positive; Test type: Other — Difference in percentage and 95% CI are based on unconditional and asymptotic Miettinen and Nurminen method; Percent Difference = -3.0, 95% CI 2-sided [-9.0 to 1.9] — Relebactam minus Placebo
Statistical Analysis 9: Comparison: Relebactam 250 mg With Imipenem/Cilastatin vs Relebactam Placebo With Imipenem/Cilastatin; Percent Diff in Participants with AEs with Rate ≥4: Headache; Test type: Other — Difference in percentage and 95% CI are based on unconditional and asymptotic Miettinen and Nurminen method; Percent Difference = 3.1, 95% CI 2-sided [-3.7 to 10.4] — Relebactam minus Placebo
Statistical Analysis 10: Comparison: Relebactam 125 mg With Imipenem/Cilastatin vs Relebactam Placebo With Imipenem/Cilastatin; Percent Diff in Participants with AEs with Rate ≥4: Headache; Test type: Other — Difference in percentage and 95% CI are based on unconditional and asymptotic Miettinen and Nurminen method; Percent Difference = -1.0, 95% CI 2-sided [-7.2 to 5.1] — Relebactam minus Placebo

11. Secondary Outcome: Percentage of Participants With a Favorable Microbiological Response at Completion of IV Study Therapy Who Had Imipenem-resistant, Gram-negative cUTI Infections.
Description: Microbiological response was assessed based on results of bacterial cultures obtained at completion of IV study medication relative to cultures obtained at baseline. A favorable microbiological response was defined as eradication of all pathogens identified at baseline. Microbiological response was assessed separately for each participant and pathogen identified in the Microbiologically Evaluable (ME) population that included participants with a urine culture confirmed to be positive for imipenem-resistant gram-negative or anaerobic infections at baseline. The overall microbiological response was determined as "favorable" if all pathogens isolated from a participant at baseline demonstrated a "favorable" response (eradication) at the time point evaluated.
Time Frame: At time of last IV dose of study drug (up to post-randomization day 14)
Population: All participants in the ME population with imipenem-resistant gram-negative infections at baseline.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Relebactam 250 mg With Imipenem/Cilastatin | Relebactam 125 mg With Imipenem/Cilastatin | Relebactam Placebo With Imipenem/Cilastatin
Number analyzed (Participants) | 10 | 7 | 6
Percentage of participants | 100.0 [69.2 to 100.0] | 100.0 [59.0 to 100.0] | 100.0 [54.1 to 100.0]

12. Secondary Outcome: Percentage of Participants With a Favorable Microbiological Response at Early Follow-up
Description: Microbiological response was assessed based on results of bacterial cultures obtained up to 9 days following completion of all study medication (IV and oral) relative to cultures obtained at baseline. A favorable microbiological response was defined as eradication of all pathogens identified at baseline. Microbiological response was assessed separately for each participant and pathogen identified in the ME population that included participants with a urine culture confirmed to be positive for at least 1 gram-negative and/or anaerobic pathogen(s) commonly isolated in UTI. The overall microbiological response was determined as "favorable" if all pathogens isolated from a participant at baseline demonstrated a "favorable" response (eradication) at the time point evaluated.
Time Frame: Up to 9 days following completion of all study IV and oral therapy (up to Day 23)
Population: All participants in the ME population with non-missing/non-indeterminate response.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Relebactam 250 mg With Imipenem/Cilastatin | Relebactam 125 mg With Imipenem/Cilastatin | Relebactam Placebo With Imipenem/Cilastatin
Number analyzed (Participants) | 65 | 72 | 71
Percentage of participants | 61.5 [48.6 to 73.3] | 68.1 [56.0 to 78.6] | 70.4 [58.4 to 80.7]

13. Secondary Outcome: Percentage of Participants With a Favorable Clinical Response at Completion of IV Study Therapy
Description: Clinical response was assessed as favorable (cured or improved) or unfavorable (failure) relative to baseline. Response determination was based on physical findings including fever (or history of fever), chills or rigors (accompanied by fever), flank pain, costovertebral angle tenderness, dysuria, urinary urgency, urinary frequency, suprapubic or pelvic pain, nausea, or vomiting. Clinical response was assessed in the ME population that included participants with a urine culture confirmed to be positive for at least 1 gram-negative and/or anaerobic pathogen(s) commonly isolated in UTI.
Time Frame: At time of last IV dose of study drug (up to postrandomization day 14)
Population: All participants in the ME population with non-missing/nonindeterminate response.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Relebactam 250 mg With Imipenem/Cilastatin | Relebactam 125 mg With Imipenem/Cilastatin | Relebactam Placebo With Imipenem/Cilastatin
Number analyzed (Participants) | 69 | 78 | 80
Percentage of participants | 97.1 [89.9 to 99.6] | 98.7 [93.1 to 100.0] | 98.8 [93.2 to 100.0]

14. Secondary Outcome: Percentage of Participants With a Favorable Clinical Response at Early Follow-up
Description: as for outcome 13
Time Frame: Up to 9 days following completion of all study IV and oral therapy (up to Day 23)
Population: All participants in the ME population with non-missing/non-indeterminate response.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Relebactam 250 mg With Imipenem/Cilastatin | Relebactam 125 mg With Imipenem/Cilastatin | Relebactam Placebo With Imipenem/Cilastatin
Number analyzed (Participants) | 64 | 73 | 76
Percentage of Participants | 89.1 [78.8 to 95.5] | 91.8 [83.0 to 96.9] | 93.4 [85.3 to 97.8]

15. Secondary Outcome: Percentage of Participants With a Favorable Clinical Response at Late Follow-up
Description: as for outcome 13
Time Frame: Up to 42 days following completion of all study IV and oral therapy (up to Day 56)
Population: All participants in the ME population with non-missing/non-indeterminate response.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Relebactam 250 mg With Imipenem/Cilastatin | Relebactam 125 mg With Imipenem/Cilastatin | Relebactam Placebo With Imipenem/Cilastatin
Number analyzed (Participants) | 62 | 71 | 76
Percentage of participants | 88.7 [78.1 to 95.3] | 87.3 [77.3 to 94.0] | 88.2 [78.7 to 94.4]

16. Secondary Outcome: Percentage of Participants With a Favorable Microbiological Response at Late Follow-up
Description: Microbiological response was assessed based on results of bacterial cultures obtained up to 42 days following completion of all study medication (IV and oral) relative to cultures obtained at baseline. A favorable microbiological response was defined as eradication of all pathogens identified at baseline. Microbiological response was assessed separately for each participant and pathogen identified in the ME population that included participants with a urine culture confirmed to be positive for at least 1 gram-negative and/or anaerobic pathogen(s) commonly isolated in UTI. The overall microbiological response was determined as "favorable" if all pathogens isolated from a participant at baseline demonstrated a "favorable" response (eradication) at the time point evaluated.
Time Frame: Up to 42 days following completion of all study IV and oral therapy (up to Day 56)
Population: All participants in the ME population with non-missing/non-indeterminate response.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Relebactam 250 mg With Imipenem/Cilastatin | Relebactam 125 mg With Imipenem/Cilastatin | Relebactam Placebo With Imipenem/Cilastatin
Number analyzed (Participants) | 63 | 69 | 72
Percentage of participants | 68.3 [55.3 to 79.4] | 65.2 [52.8 to 76.3] | 62.5 [50.3 to 73.6]

ADVERSE EVENTS:
Time Frame: Up to 42 days following completion of all study therapy for drug-related serious adverse events (up to 56 days); and up to 14 days following completion of all study therapy for all-cause serious and non-serious adverse events (up to 28 days).
Description: AEs were reported for the All Participants as Treated Population that included all randomized participants who received ≥ 1 dose of study treatment. All-Cause Mortality included deaths outside the 14 day follow up period.
Arm/Group | Relebactam 250 mg With Imipenem/Cilastatin | Relebactam 125 mg With Imipenem/Cilastatin | Relebactam Placebo With Imipenem/Cilastatin
All-Cause Mortality (participants affected / at risk) | 2/99 | 0/99 | 0/100
Serious Adverse Events (participants affected / at risk) | 5/99 | 2/99 | 3/100
Other Adverse Events (participants affected / at risk) | 11/99 | 9/99 | 7/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Relebactam 250 mg With Imipenem/Cilastatin (N=99) | Relebactam 125 mg With Imipenem/Cilastatin (N=99) | Relebactam Placebo With Imipenem/Cilastatin (N=100)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Glomerulonephritis rapidly progressive (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Relebactam 250 mg With Imipenem/Cilastatin (N=99) | Relebactam 125 mg With Imipenem/Cilastatin (N=99) | Relebactam Placebo With Imipenem/Cilastatin (N=100)
Headache (Nervous system disorders) | 7 (7) | 3 (3) | 4 (4)
Nausea (Gastrointestinal disorders) | 4 (4) | 6 (6) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission.